CLINICAL TRIAL: NCT04752969
Title: Can Thyroid Levels Affect Topographic, Densitometric and Aberrometric Values of the Cornea
Brief Title: The Effect of Thyroid Hormon Levels on the Corneal Measures
Status: Completed | Type: Observational
Sponsor: Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Mehmet Fuat Alakuş, assistant professor, Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital
Other Study IDs: 30012021
Record Dates: First submitted 2021-01-31; First posted 2021-02-12 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Thyroid Disorder; Corneal Opacity
Keywords: Thyroid disorder; Corneal opacity; Corneal aberrations
MeSH Terms: conditions — Thyroid Diseases; Corneal Opacity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Hypothyroidia: 20 subjects diagnosed with hypothyroidism
- Hyperthyroidia: 20 subjects diagnosed with hyperthyroidism
- Healthy: 20 age-matched healthy control subjects

SUMMARY:
In this cross-sectional comparative study, it is aimed to investigate the topographic measurements,aberrometrics and densitometrics values of corneas in hypothyroid and hyperthyroid patients compared to healthy individuals. A number of 20 hypothyroid patients (group I), 20 hyperthyroid patients (group II), and 20 age-matched healthy controls (group III) have been recruited. The Pentacam high resolution imaging system is used to determine corneal topographic measurements,aberrometry and densitometry.

DETAILED DESCRIPTION:
Thyroid hormone diseases can cause different symptoms and signs in the body according to the hormone levels, particularly in the eyes. Corneal tissue can be affected by many biochemical and hormonal factors, and many ocular surface and systemic diseases can affect the cornea.Hyperthyroidism has been shown to cause symptoms such as conjunctival chemosis, proptosis, increased intraocular pressure, limitation to globe movements due to the restriction of extraocular muscles, increased orbital volume, increased risk of glaucoma with inflammation in the trabecular meshwork and exposure keratopathy, especially in Graves' disease. In the case of hypothyroidism, studies have shown fluid retention and edema in all body tissues, thereby resulting in increased thickness in the cornea, as well as a decrease in corneal hysteresis, which increases the risk of glaucoma. In this study, it is aimed to assess whether thyroid hormone changes affect those parameters by objectively measuring corneal changes via corneal topography, corneal densitometry and corneal aberrometry.

ELIGIBILITY:
Inclusion Criteria:

* Thyroid hormone disorder patients with a novel diagnosis
* Age-matched healthy individuals without any systemic disorder (e.g., diabetes mellitus, hypertension, rhematoid artritis, asthma etc.)

Exclusion Criteria:

* Having a spherical or cylindrical refractive error of >1.0 degrees,
* Congenital corneal dystrophies, corneal ectasia, corneal ulcers or scars, keratitis, ocular surface infections, keratoconus,
* A history of ocular trauma,
* Uveitis,
* Glaucoma,
* A history of contact lens wear,
* A history of ocular surgery,
* Dry eye diseases

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 20 patients diagnosed hypthyroidia ,20 patients diagnosed hyperthyroidia ,20 age matched healthy individuals
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
corneal density in throid patients | up to 12 weeks
  corneal density values according to type of thyroid disorder

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet F Alakuş, MD, Principal Investigator — Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital
Locations (1):
- Sağlık Bilimleri Üniversitesi Gazi Yaşargil Training and Research Hospital, Diyarbakır, Turkey (Türkiye)

REFERENCES:
- [Result] Cankurtaran V, Tekin K, Cakmak AI, Inanc M, Turgut FH. Assessment of corneal topographic, tomographic, densitometric, and biomechanical properties of Fabry patients with ocular manifestations. Graefes Arch Clin Exp Ophthalmol. 2020 May;258(5):1057-1064. doi: 10.1007/s00417-019-04593-8. Epub 2020 Jan 8. PMID 31915973
- [Result] Bilgihan K, Hondur A, Sul S, Ozturk S. Pregnancy-induced progression of keratoconus. Cornea. 2011 Sep;30(9):991-4. doi: 10.1097/ICO.0b013e3182068adc. PMID 21705880
- [Result] Villani E, Viola F, Sala R, Salvi M, Mapelli C, Curro N, Vannucchi G, Beck-Peccoz P, Ratiglia R. Corneal involvement in Graves' orbitopathy: an in vivo confocal study. Invest Ophthalmol Vis Sci. 2010 Sep;51(9):4574-8. doi: 10.1167/iovs.10-5380. Epub 2010 Apr 30. PMID 20435595